CLINICAL TRIAL: NCT00239278
Title: Effects of High Dose Inhaled Budesonide+ Formoterol Versus Placebo and Oral Prednisolone on Biomarkers of Airway Inflammation in the Treatment of Exacerbations in Non-hospitalised Patients With Mild to Moderate COPD.
Brief Title: Budesonide / Formoterol in Treatment of Exacerbations of COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-039-0698; D5892C00698 (Other: AstraZeneca)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination; Prednisolone

INTERVENTIONS:
Drug: budesonide/formoterol, 2x 200/6 microgram. 4 times daily
  Other Names: Symbicort
Drug: prednisolone, 30 mg once daily and placebo

SUMMARY:
The purpose of this study is to determine whether the budesonide+formoterol combination is effective in the treatment of exacerbations of COPD with a main emphasis on investigating the effects on inflammation and a secondary emphasis on clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

* smoking-induced COPD according to ATS criteria
* FEV1 <85% of predicted at enrolment and <70% of predicted but > 0.7 Liter at Exacerbation
* FEV1/IVC ratio <88% of predicted for men and <89% for women

Exclusion Criteria:

* history of asthma
* known hypersensitivity to the study drugs
* serious concomitant diseases
* pregnancy or lactating
* abnormal Chest X-ray or blood gasses

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-01; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Eosinophils in induced sputum (as % of Total Cell Count), change from the start of the exacerbation to the end of 14 days treatment

SECONDARY OUTCOMES:
Inflammatory markers in induced sputum, blood/serum and urine
Lung function tests at clinic
Diary cards for PEF and symptoms
Patient Related outcomes
Questioning for Adverse Events and in blood: routine tests and cortisol

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Groningen, Netherlands

REFERENCES:
- [Derived] Bathoorn E, Liesker JJ, Postma DS, Boorsma M, Bondesson E, Koeter GH, Kauffman HF, van Oosterhout AJ, Kerstjens HA. Anti-inflammatory effects of combined budesonide/formoterol in COPD exacerbations. COPD. 2008 Oct;5(5):282-90. doi: 10.1080/15412550802363360. PMID 18972276
- [Derived] Bathoorn E, Liesker J, Postma D, Koeter G, van Oosterhout AJ, Kerstjens HA. Safety of sputum induction during exacerbations of COPD. Chest. 2007 Feb;131(2):432-8. doi: 10.1378/chest.06-2216. PMID 17296644